CLINICAL TRIAL: NCT06826144
Title: Chronic Remote Ischemic Conditioning in Small Infarctions Associated with Stent-assisted Coiling of Unruptured Intracranial Aneurysms: a Single-center Randomized Controlled Trial.
Brief Title: Chronic Remote Ischemic Conditioning in Small Infarctions Associated with Stent-assisted Coiling of Unruptured Intracranial Aneurysms
Acronym: CRISIS
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The First Affiliated Hospital with Nanjing Medical University (Other)
Responsible Party: Principal Investigator, Lu Hua, professor, The First Affiliated Hospital with Nanjing Medical University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: CRISIS
Record Dates: First submitted 2025-02-10; First posted 2025-02-13 (Actual); Last update posted 2025-02-13 (Actual); Status verified 2025-01

CONDITIONS: Unruptured Intracranial Aneurysm; Infarction Cerebral
Keywords: remote ischemic conditioning
MeSH Terms: conditions — Cerebral Infarction

STUDY DESIGN:
Intervention Model Description: Standard Treatment All enrolled patients receive standard stent-assisted aneurysm coiling therapy. Depending on intraoperative and postoperative conditions, tirofiban is administered as follows: an initial bolus of 0.6 μg/kg over 3 minutes, followed by continuous intravenous infusion at 0.1 μg/kg/min for 18 hours.
  RIC Treatment Protocol Remote ischemic conditioning (RIC) is applied to the contralateral upper limb, consisting of 5 cycles per session, 2 sessions per day. Each cycle includes 5 minutes of ischemia followed by 5 minutes of reperfusion. The pressure used to occlude the brachial artery is set at 200 mmHg or exceeds baseline systolic pressure by 35 mmHg (intervention group) or 20 mmHg (control group).
  Group Assignments
  Group A (Control Group):
  At least 4 sessions of sham RIC treatment before the procedure. Continued sham RIC treatment for a minimum of 4 weeks postoperatively.
  Group B (Intervention Group):
  At least 4 sessions of actual RIC treatment before the procedure. Cont
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- RIC (Experimental): All enrolled patients receive standard stent-assisted aneurysm coiling therapy（Patients are required to receive antiplatelet therapy for at least 3 days before the procedure, consisting of:Aspirin: 100 mg once daily, combined with Clopidogrel: 75 mg once daily, or Ticagrelor: 90 mg twice daily）.Depending on intraoperative and postoperative conditions, tirofiban is administered as follows: an initial bolus of 0.6 μg/kg over 3 minutes, followed by continuous intravenous infusion at 0.1 μg/kg/min for 18 hours.
  Remote ischemic conditioning (RIC) is applied to the contralateral upper limb, consisting of 5 cycles per session, 2 sessions per day. Each cycle includes 5 minutes of ischemia followed by 5 minutes of reperfusion. The pressure used to occlude the brachial artery is set at 200 mmHg or exceeds baseline systolic pressure by 35 mmHg At least 4 sessions of actual RIC treatment before the procedure.Continued RIC treatment for a minimum of 4 weeks postoperatively.
  Interventions: Procedure: remote ischemic conditioning
- sham (Sham Comparator): All enrolled patients receive standard stent-assisted aneurysm coiling therapy.（Patients are required to receive antiplatelet therapy for at least 3 days before the procedure, consisting of:Aspirin: 100 mg once daily, combined with Clopidogrel: 75 mg once daily, or Ticagrelor: 90 mg twice daily）.Depending on intraoperative and postoperative conditions, tirofiban is administered as follows: an initial bolus of 0.6 μg/kg over 3 minutes, followed by continuous intravenous infusion at 0.1 μg/kg/min for 18 hours.
  Remote ischemic conditioning (RIC) is applied to the contralateral upper limb, consisting of 5 cycles per session, 2 sessions per day. Each cycle includes 5 minutes of ischemia followed by 5 minutes of reperfusion. The pressure used to occlude the brachial artery is set at 20 mmHg.
  At least 4 sessions of sham RIC treatment before the procedure.Continued sham RIC treatment for a minimum of 4 weeks postoperatively.
  Interventions: Procedure: Sham treatment

INTERVENTIONS:
Procedure: remote ischemic conditioning — Remote ischemic conditioning (RIC) is applied to the contralateral upper limb, consisting of 5 cycles per session, 2 sessions per day. Each cycle includes 5 minutes of ischemia followed by 5 minutes of reperfusion. The pressure used to occlude the brachial artery is set at 200 mmHg or exceeds baseline systolic pressure by 35 mmHg (intervention group).At least 4 sessions of actual RIC treatment before the procedure.Continued RIC treatment for a minimum of 4 weeks postoperatively.
  Other Names: RIC
  Arms: RIC
Procedure: Sham treatment — Remote ischemic conditioning (RIC) is applied to the contralateral upper limb, consisting of 5 cycles per session, 2 sessions per day. Each cycle includes 5 minutes of ischemia followed by 5 minutes of reperfusion. The pressure used to occlude the brachial artery is set at 20 mmHg.At least 4 sessions of sham RIC treatment before the procedure.Continued sham RIC treatment for a minimum of 4 weeks postoperatively.
  Arms: sham

SUMMARY:
1. Disease Description Stent-assisted coiling has become an effective treatment modality for intracranial aneurysms. With continuous advancements in periprocedural antiplatelet regimens, the incidence of symptomatic thromboembolic events has significantly decreased. However, the rate of procedure-related microembolic infarctions, which are characterized by punctate hyperintense signals on DWI, remains high (10%-76.5%). The underlying causes of these microembolic infarctions remain controversial and may be associated with factors such as different stent types, sheath types, antiplatelet regimens, intraoperative adverse events (e.g., vascular dissection or spasm), patient age, and procedure duration. While most patients with microembolic infarctions exhibit no overt clinical symptoms, the presence of these infarctions reflects underlying tissue damage, posing potential risks that cannot be ignored. Furthermore, their occurrence highlights insufficient preoperative preparation or intraoperative technical issues, which may increase the likelihood of symptomatic embolism. Therefore, investigating the causes of microembolic infarctions and exploring preventive strategies is of great clinical significance.
2. Intervention Description Remote ischemic conditioning (RIC) involves inducing temporary ischemia in distal vessels to protect target vessels from ischemic and reperfusion injuries. RIC can be performed before, during, or after ischemic events and is widely used in the context of coronary artery ischemia. Some studies have shown that RIC can mitigate ischemia-related injuries in the myocardium, kidneys, and lower limbs following cardiovascular surgeries. Previous research has also demonstrated the neuroprotective effects of RIC in ischemia-reperfusion injuries of the nervous system. For instance, RIC significantly improves outcomes in cerebral small vessel disease (CSVD)-related acute stroke events and ameliorates cognitive impairments associated with CSVD. Moreover, the safety and efficacy of RIC have been validated in other conditions or procedures, such as aneurysmal subarachnoid hemorrhage (aSAH), intracranial atherosclerotic stenosis, and carotid artery stenting.
3. Research Hypothesis Current clinical studies on RIC have primarily focused on acute ischemic stroke (including large artery atherosclerosis and CSVD), spontaneous intracerebral hemorrhage, and subarachnoid hemorrhage. The Remote Ischemic Conditioning for Acute Stroke Trial (RESIST) indicated that RIC effectively improves outcomes in acute strokes related to CSVD, including reducing white matter hyperintensities, infarct volume, and modified Rankin Scale (mRS) scores. A clinical study conducted at the Mayo Clinic demonstrated the safety of remote ischemic preconditioning (RIPC) during intracranial aneurysm coiling. Our center's previous study on "Tirofiban and Procedure-Related Microemboli in Stent-Assisted Aneurysm Coiling" revealed that the incidence of procedure-related microembolic infarctions was 61.1% in the non-tirofiban group and 19.4% in the tirofiban-treated group. However, there is currently a lack of research on the use of RIC for procedure-related microembolic infarctions in stent-assisted aneurysm coiling.

This study aims to explore the efficacy of ischemic conditioning treatment, performed preoperatively and postoperatively, in reducing procedure-related microembolic infarctions during standard stent-assisted aneurysm coiling. The primary outcomes include the incidence of acute microembolic infarctions postoperatively and the incidence of symptomatic microembolic infarctions at one month following RIC.

ELIGIBILITY:
Inclusion Criteria:

* 1) Age 18-80; 2) Unruptured aneurysm with surgical indications; 3) Stent assisted aneurysm embolization; 4) Patients were willing to receive ischemic adaptation therapy.

Exclusion Criteria:

* 1) Age < 18 years old; 2) Complicated with cerebrovascular malformations, moyamoya disease and other hemorrhagic cerebrovascular diseases or history; 3) pregnancy; 4) History of acute myocardial infarction within 1 month; 5) Peripheral vascular disease or peripheral neuropathy of the upper limb; 6) Upper limb vascular and soft tissue injury, or combined with limb deformity; 7) Severe subclavian artery stenosis or occlusion; 8) Poor blood pressure control, upper extremity basal systolic pressure ≥200mmHg; 9) Chronic kidney disease.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Estimated)
Dates: Start 2025-02-20 (Estimated); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
Efficacy of Remote Ischemic Conditioning (RIC) in Preventing Small Infarctions Associated with Stent-Assisted Aneurysm Coiling | Within 24 hours after the procedure,
  Within 24 hours after the procedure, a brain MRI is performed to record the number and size of hyperintense signals on DWI. The trial group and control group are compared, and the efficacy is assessed based on statistical analysis results. If the mean number of hyperintense signals on DWI in the trial group is lower than that in the control group, with a statistically significant difference, the intervention is considered effective; otherwise, it is considered ineffective.

SECONDARY OUTCOMES:
Efficacy of Chronic Remote Ischemic Conditioning (RIC) in Treating Small Infarctions Associated with Stent-Assisted Aneurysm Coiling | One month after the procedure
  One month after the procedure, a follow-up brain MRI is performed to evaluate the infarct area and number based on the size and number of hyperintense signals observed on DWI at 24 hours postoperatively. Additionally, the modified Rankin Scale (mRS) is completed one month postoperatively. The trial group and control group are compared, and efficacy is assessed based on statistical analysis results. If the mean infarct area and number in the trial group are lower than those in the control group, with statistically significant differences, the intervention is considered effective; otherwise, it is deemed ineffective. Similarly, if the mRS score distribution in the trial group is lower than that in the control group, with statistically significant differences, the intervention is considered effective; otherwise, it is considered ineffective.

OTHER OUTCOMES:
The incidence of thrombus formation or embolic events in the limb subjected to RIC in the intervention group. | 24 hours, 2 weeks, and 1 month postoperatively
  Vascular ultrasound of the limb subjected to RIC will be performed at 24 hours, 2 weeks, and 1 month postoperatively to assess for thrombus formation or thromboembolism.
The incidence of skin damage or bruising in the RIC group. | before surgery and 24 hours, 2 weeks, and 1 month postoperatively

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Mohammad Seyedsaadat S, Rangel Castilla L, Lanzino G, Cloft HJ, Blezek DJ, Theiler A, Kadirvel R, Brinjikji W, Kallmes DF. Remote ischemic preconditioning for elective endovascular intracranial aneurysm repair: a feasibility study. Neuroradiol J. 2019 Jun;32(3):166-172. doi: 10.1177/1971400919842059. Epub 2019 Apr 3. PMID 30942660
- [Background] Zhao W, Meng R, Ma C, Hou B, Jiao L, Zhu F, Wu W, Shi J, Duan Y, Zhang R, Zhang J, Sun Y, Zhang H, Ling F, Wang Y, Feng W, Ding Y, Ovbiagele B, Ji X. Safety and Efficacy of Remote Ischemic Preconditioning in Patients With Severe Carotid Artery Stenosis Before Carotid Artery Stenting: A Proof-of-Concept, Randomized Controlled Trial. Circulation. 2017 Apr 4;135(14):1325-1335. doi: 10.1161/CIRCULATIONAHA.116.024807. Epub 2017 Feb 7. PMID 28174194
- [Background] Meng R, Ding Y, Asmaro K, Brogan D, Meng L, Sui M, Shi J, Duan Y, Sun Z, Yu Y, Jia J, Ji X. Ischemic Conditioning Is Safe and Effective for Octo- and Nonagenarians in Stroke Prevention and Treatment. Neurotherapeutics. 2015 Jul;12(3):667-77. doi: 10.1007/s13311-015-0358-6. PMID 25956401
- [Background] Laiwalla AN, Ooi YC, Liou R, Gonzalez NR. Matched Cohort Analysis of the Effects of Limb Remote Ischemic Conditioning in Patients with Aneurysmal Subarachnoid Hemorrhage. Transl Stroke Res. 2016 Feb;7(1):42-8. doi: 10.1007/s12975-015-0437-3. Epub 2015 Dec 2. PMID 26630942
- [Background] Wang Y, Meng R, Song H, Liu G, Hua Y, Cui D, Zheng L, Feng W, Liebeskind DS, Fisher M, Ji X. Remote Ischemic Conditioning May Improve Outcomes of Patients With Cerebral Small-Vessel Disease. Stroke. 2017 Nov;48(11):3064-3072. doi: 10.1161/STROKEAHA.117.017691. Epub 2017 Oct 17. PMID 29042490
- [Background] Blauenfeldt RA, Mortensen JK, Hjort N, Valentin JB, Homburg AM, Modrau B, Sandal BF, Gude MF, Berhndtz AB, Johnsen SP, Hess DC, Simonsen CZ, Andersen G. Effect of Remote Ischemic Conditioning in Ischemic Stroke Subtypes: A Post Hoc Subgroup Analysis From the RESIST Trial. Stroke. 2024 Apr;55(4):874-879. doi: 10.1161/STROKEAHA.123.046144. Epub 2024 Feb 1. PMID 38299363
- [Background] Eitel I, Stiermaier T, Rommel KP, Fuernau G, Sandri M, Mangner N, Linke A, Erbs S, Lurz P, Boudriot E, Mende M, Desch S, Schuler G, Thiele H. Cardioprotection by combined intrahospital remote ischaemic perconditioning and postconditioning in ST-elevation myocardial infarction: the randomized LIPSIA CONDITIONING trial. Eur Heart J. 2015 Nov 21;36(44):3049-57. doi: 10.1093/eurheartj/ehv463. Epub 2015 Sep 17. PMID 26385956
- [Background] Luo SJ, Zhou YJ, Shi DM, Ge HL, Wang JL, Liu RF. Remote ischemic preconditioning reduces myocardial injury in patients undergoing coronary stent implantation. Can J Cardiol. 2013 Sep;29(9):1084-9. doi: 10.1016/j.cjca.2012.11.022. Epub 2013 Feb 12. PMID 23414904
- [Background] Hausenloy DJ, Yellon DM. Remote ischaemic preconditioning: underlying mechanisms and clinical application. Cardiovasc Res. 2008 Aug 1;79(3):377-86. doi: 10.1093/cvr/cvn114. Epub 2008 May 2. PMID 18456674
- [Background] Bell R, Yellon D. Surgery: Remote ischaemic conditioning--approaching prime time? Nat Rev Cardiol. 2013 Nov;10(11):619-21. doi: 10.1038/nrcardio.2013.154. Epub 2013 Sep 24. No abstract available. PMID 24060957
- [Background] Kim DY, Park JC, Kim JK, Sung YS, Park ES, Kwak JH, Choi CG, Lee DH. Microembolism after Endovascular Treatment of Unruptured Cerebral Aneurysms: Reduction of its Incidence by Microcatheter Lumen Aspiration. Neurointervention. 2015 Sep;10(2):67-73. doi: 10.5469/neuroint.2015.10.2.67. Epub 2015 Sep 2. PMID 26389009
- [Background] Park JC, Lee DH, Kim JK, Ahn JS, Kwun BD, Kim DY, Choi CG. Microembolism after endovascular coiling of unruptured cerebral aneurysms: incidence and risk factors. J Neurosurg. 2016 Mar;124(3):777-83. doi: 10.3171/2015.3.JNS142835. Epub 2015 Sep 18. PMID 26381257
- [Background] Bendszus M, Koltzenburg M, Burger R, Warmuth-Metz M, Hofmann E, Solymosi L. Silent embolism in diagnostic cerebral angiography and neurointerventional procedures: a prospective study. Lancet. 1999 Nov 6;354(9190):1594-7. doi: 10.1016/S0140-6736(99)07083-X. PMID 10560674